CLINICAL TRIAL: NCT06781840
Title: The Feasibility of the Promoting Health Through Play Opportunities Program in Improving Parent and Child Outcomes for Underserved Families.
Brief Title: Promoting Health Through Play Program: Improving Parent and Child Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Collaborators: Head Start (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20226278
Record Dates: First submitted 2024-09-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-08

CONDITIONS: Child Development; Parenting
Keywords: play; playfulness; parent-group educational training

STUDY DESIGN:
Intervention Model Description: 2 groups: One for English speaking parents and the other for Spanish speaking parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Promoting Health Through Play English version (Experimental): Parent online group sessions- English version consisting of five 45-minute-long parent group online sessions. In addition, each parent-child dyad will receive, one 30-minute-long online guided play session with OTS/OT.
  Interventions: Behavioral: Playing Playfully to Overcome Adversity
- Promoting Health Through Play Spanish version (Other): Parent online group sessions- Spanish version consisting of five 45-minute-long parent group online sessions. In addition, each parent-child dyad will receive, one 30-minute-long online guided play session with OTS/OT.
  Interventions: Behavioral: Playing Playfully to Overcome Adversity

INTERVENTIONS:
Behavioral: Playing Playfully to Overcome Adversity — The intervention will consist of two parts: (a) five 45-minute-long parent group online sessions; and (b) one 30-minute long online guided play session with OTS/OT.The training will consist of asynchronous module and PowerPoint presentations followed by role play and discussions.
  Other Names: Promoting Health Through Play Opportunities program

SUMMARY:
This project aims to assess the feasibility of an intervention program consisting of parent online group sessions in addition to guided individual play session between parent, child, and occupational therapy student (OTS) or an occupational therapist (OT).

The investigators speculate that the Promoting Health Through Play Opportunities program will be effective in improving:

1. Parent ability to support their child's playfulness as measured during 15-minute video-recorded joint play activity at home using the Parent/Caregiver Support of Childre Playfulness [PC-SCP].
2. Child's playfulness behavior as measured during 15-minute video-recorded joint play activity at home using the Test of Playfulness [ToP].
3. Child's psychological adjustment as measured by the Strength and Difficulties Questionnaire [SDQ].
4. Parent's perception and satisfaction from their involvement in the program as measured through open-ended questions.

DETAILED DESCRIPTION:
The Promoting Health Through Play Opportunities program (Halperin et al., 2021; Waldman-Levi & Halperin, 2022) is a strength-based intervention that provides tools to help parents become change agents in their child's life through the promotion of healthy play opportunities within the family context. This research project aims to enhance children's development through playful interactions with their parents. The investigators speculate that the program will be effective in improving parent and child joint play experience and child's social-emotional functioning.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Head Start pre-school program within New York greater area
* Parent-child dyads
* Child must be 3 to 5 years old, with/without delay or disability.
* If a parent has more than one child in this age range, the oldest of them will be recruited for the study
* Parent IS committed to attending pre-and-posttest as well as online group sessions
* Parent has access to a device other than a phone (tablet, iPad, laptop) and has stable internet connection to be able to participate in the online group and dyadic session
* For the English-speaking group, parent must be fluent in English
* For the Spanish speaking group, parent must be fluent in the Spanish language.

Exclusion Criteria:

* Parents with a sensory deficit (e.g., hearing or vision impairment) that will affect their ability to participate in an online group program
* Parents with psychiatric or behavioral disorders that affect their ability to participate in a group-based intervention

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire. Goodman R. (1997). The Strengths and Difficulties Questionnaire: A research note. 38(5), 581-586. doi:10.1111/j.1469-7610.1997.tb01545.x | through study completion, an average of 6 weeks
  The Strengths and Difficulties Questionnaire assesses child's psychological adjustment. It contains 25 items measured on a scale ranging from 0 (no difficulty) to 2 (severe difficulty).
Parent/Caregiver Support of Children Playfulness (PC-SCP). Waldman-Levi, A., & Bundy, A. (2023). Parent/Caregiver Support of Children Playfulness (PC-SCP). AOTA Press. | through study completion, an average of 6 weeks
  The PC-SCP assesses how parents or primary caregivers support children's ability to play. It is based on a 15-minute video-recorded observation of a parent-child joint play and contains 16 items. Scores range from 0 (low level of parent support of child's play or playfulness) to 3 (high level of parent support of child's play or playfulness).
Test of Playfulness. Skard, G., & Bundy, A. C. (2008). Test of Playfulness. In L. D. Parham &amp; L. S. Fazio (Eds.), Play in occupational therapy for children (2nd ed., pp. 71-93). St. Louis, MO: Mosby, Inc | through study completion, an average of 6 weeks
  The ToP assesses children's ability to play in a playful manner. It is observed during video-recorded 15-minute play and contains 30 items. Scores range from 0 (low level of child's playfulness behavior) to 3 (high level of child's playfulness behavior).

SECONDARY OUTCOMES:
Parent post program interview | 6 weeks
  Semi-structured recorded interview

CONTACTS AND LOCATIONS:
Locations (1):
- Head Start, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No